CLINICAL TRIAL: NCT05186727
Title: You Cannot Change Your Family History, But You Can Change What You do With it: A Peer-based Education Program to Reduce Breast Cancer Risk in African American Women
Brief Title: Family History and Breast Cancer Education Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Laurene Tumiel Berhalter, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00005038
Record Dates: First submitted 2021-11-06; First posted 2022-01-11 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Genetic Predisposition to Disease
Keywords: Family History; African American; Breast Cancer Screening
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Researcher-Group (Active Comparator): Education delivered in a group session by a member of the research team
  Interventions: Other: Family History education
- Research-One on One (Active Comparator): Education delivered telephonically one-on-one by a member of the research team
  Interventions: Other: Family History education
- Patient Ambassador-Group (Active Comparator): Education delivered in a group session by a Patient Ambassador (a peer mentor)
  Interventions: Other: Family History education; Other: Patient Ambassador
- Patient Ambassador- One on One (Active Comparator): Education delivered telephonically one-on-one by a Patient Ambassador (peer mentor)
  Interventions: Other: Family History education; Other: Patient Ambassador

INTERVENTIONS:
Other: Family History education — The education, developed in partnership with community partners, intends to assist women to collect family history of breast cancer and share it with their providers.
Other: Patient Ambassador — The support of a Patient Ambassador in addition to the education is also tested.
  Arms: Patient Ambassador- One on One; Patient Ambassador-Group

SUMMARY:
The overall goal of this study is to reduce breast cancer morbidity and mortality disparities among African American women by actively engaging family history as a tool to modify screening regimens and enhance communication between women and their providers. Therefore, this rationale is reflected the project title: "You cannot change your family history, but you can change what you do with it: A peer-based education program to reduce breast cancer risk in African American women"

This study will develop and test an educational curriculum that highlights the importance of knowing family history and sharing it with health care providers. The curriculum will include tools to gather family history and discuss it with providers to guide the delivery of care. The investigators will assess the effectiveness of the curriculum in group and one-on-one settings and when delivered by a Patient Ambassador (peer train-the trainer model) or a researcher.

The specific objectives of the study are to:

Obj. 1: Develop a CBPR-based curriculum- using a community based participatory research (CBPR) approach, that highlights the importance of family history as a risk factor for breast cancer that includes tools to collect family history information and discuss it with providers to enable a family history based screening regimen.

Obj. 2: Train Patient Ambassadors- Patient Ambassadors, women from the community who act as community messengers to deliver the curriculum.

Obj. 3: Pilot Implementation and Extensive Evaluation of the Curriculum- Assess two modes of delivery, group vs one-on-one, and Peer Ambassadors vs. a researcher.

Obj. 4: Dissemination- of the curricular products, implementation pilot results, and implementation guides for communities and practices- via publications and other channels in preparation for grant submits to enhance the program.

DETAILED DESCRIPTION:
Women from underserved communities are eligible to participate in the educational workshop and the evaluation of the study. We aim to recruit 200 women; 50 randomized into each arm (researcher group, researcher one-on-one, Patient Ambassador group, Patient Ambassador one-on-one) of the evaluation. Participants will be recruited from community-based sources such as the Buffalo Research Registry, primary care practices, and word of mouth through Patient Voices Network, Our Curls, and other community-based organizations. It is anticipated that most of these women will be African American as recruitment will be geared toward predominately African American communities. A marketing flyer, available in e-mail or print format, will be developed to disseminate through the various community-based strategies. Women will be consented and randomized telephonically. Randomization without replacement will be used for every four women consented to ensure equal groups. The research associate will conduct the baseline assessment will be collected over the telephone to maintain the evaluation separate from the implementation of the curriculum. Curriculum content areas include: Breast health knowledge, Breast cancer knowledge, Family History Genetics, Breast Cancer Genetic Testing Methods, and how to collect family history information. Women randomized into the one-on-one phone interventions will be immediately linked to either the Patient Ambassador or researcher who will be administering the curriculum. An initial contact will be made for introductions, to describe the process and schedule four additional times for phone calls. One phone call will be made per week for four weeks. A packet of materials, that include curriculum handouts and supporting tools, will be sent to the participant for follow-up calls. The Patient Ambassador or professional will then follow up with each participant according to the arranged schedule. For participants randomized to the group sessions, 4 dates will be offered at the time of consent for an average of 12-13 participants at each group. Participants will be asked to choose one date. The same materials and tools will be given to the women at the beginning of the session. The curriculum will be delivered in a more didactic approach with time for group interaction and hands on activities. The sessions will be conducted via ZOOM. A fidelity checklist will be created that a member of the research team will complete for both group sessions and will spot check 20% or the on-on-one needs to complete to ensure completion of the full curriculum and protocols is adhered to. Once a month contacts will be made by the individual that delivered the curriculum as a retention strategy. Assessments are conducted immediately after the intervention and three months after the close of the education. These surveys will consist of the same measures included in the baseline and will add a measure about satisfaction with the curriculum, the facilitator, and the mode of delivery.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age and older
* Live in predominately African American communities (ZIP codes)

Exclusion Criteria:

* No previous breast cancer diagnosis

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 196 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge of Genetic Screening for Breast Cancer | Baseline
  The breast cancer genetic counseling knowledge questionnaire will be used to assess knowledge. This tool was validated by nurses, genetic counselors, and a group of employees.
Change in Knowledge of Genetic Screening for Breast Cancer | 1 week Post Intervention
  The breast cancer genetic counseling knowledge questionnaire will be used to assess knowledge. This tool was validated by nurses, genetic counselors, and a group of employees.
Change in Knowledge of Genetic Screening for Breast Cancer | 3 Months Post Intervention
  The breast cancer genetic counseling knowledge questionnaire will be used to assess knowledge. This tool was validated by nurses, genetic counselors, and a group of employees.
Change intention to be screened and to gather family history and share with providers | Baseline
  Other items to be assessed will include attitude towards screening and family history, intent to be screened, intent to gather family history, and intent to discuss family history of breast cancer with their providers. The PRECEDE-PROCEED model will serve as a framework for the evaluation of intent to change. This model serves as a method to measure the socioecological, educational, and social epidemiological aspects of behavior change.
Change intention to be screened and to gather family history and share with providers | 1 week Post Intervention
  Other items to be assessed will include attitude towards screening and family history, intent to be screened, intent to gather family history, and intent to discuss family history of breast cancer with their providers. The PRECEDE-PROCEED model will serve as a framework for the evaluation of intent to change. This model serves as a method to measure the socioecological, educational, and social epidemiological aspects of behavior change.
Change intention to be screened and to gather family history and share with providers | 3 Months Post Intervention
  Other items to be assessed will include attitude towards screening and family history, intent to be screened, intent to gather family history, and intent to discuss family history of breast cancer with their providers. The PRECEDE-PROCEED model will serve as a framework for the evaluation of intent to change. This model serves as a method to measure the socioecological, educational, and social epidemiological aspects of behavior change.

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No